CLINICAL TRIAL: NCT00927550
Title: Randomized Evaluation of the Effectiveness of Lithium in Subjects With Treatment-Resistant Depression and Suicide Risk. An Independent, Pragmatic, Multicentre, Parallel-Group, Superiority Trial
Brief Title: Lithium and Standard Therapy in Resistant Depression
Acronym: LAST
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universita di Verona (Other)
Responsible Party: Corrado Barbui MD, University of Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAST_RD_FARM77Z3BL-5.1_132009
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Depression
Keywords: resistant depression; lithium; RCT; lithium therapy; standard therapy
MeSH Terms: conditions — Depression | interventions — Lithium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lithium plus usual care (Experimental)
  Interventions: Drug: lithium
- usual care without lithium therapy (Active Comparator)
  Interventions: Drug: usual care

INTERVENTIONS:
Drug: lithium — Patients allocated to lithium will be administered an oral starting dose ranging between 150 and 300 milligrams. Suggested final oral dose will have to achieve plasma levels of 0.4 to 1.0 mmol/L. Clinicians will be free of increasing or decreasing the dose according to clinical status and circumstances. Dose changes will be recorded. Following randomization, treatment is to be taken daily for 1 year unless some clear reason to stop develops. Patients allocated to the lithium arm will receive usual pharmacological and non-pharmacological treatment as clinically indicated. Any other pharmacological treatment will be allowed.
  Other Names: Carbolithium
  Arms: lithium plus usual care
Drug: usual care — Patients allocated to the control arm will receive usual pharmacological and non-pharmacological treatment as clinically indicated. Patients allocated to the control arm will not be allowed to receive lithium. Any other pharmacological treatment will be allowed.
  Arms: usual care without lithium therapy

SUMMARY:
The principal clinical question is whether lithium is effective in reducing the risk of suicidal behaviour in subjects with treatment-resistant depression and suicide risk. Additionally aims of the study are: (a) to assess whether lithium is effective in improving depressive symptomatology in subjects with treatment-resistant depression and suicide risk; (b) to assess the tolerability profile of lithium.

DETAILED DESCRIPTION:
Inclusion criteria:

1. Diagnosis of major depression (clinical diagnosis, guided by DSM-IV criteria).
2. History of attempted suicide or deliberate self-harm in the previous 12 months.
3. Inadequate response to at least two antidepressants given sequentially at an adequate dose for an adequate time for the current depressive episode.
4. Uncertainty about which treatment arm would be best for the participant.
5. Age 18 or above.
6. Agreement between investigator and patient to enter the study.

Exclusion criteria:

1. In addition to major depression, a primary diagnosis of any concurrent Axis I disorder (according to DSM-IV criteria) will constitute an exclusion criterion; by contrast, any concurrent Axis II disorder (according to DSM-IV criteria) will not constitute an exclusion criterion.
2. Previous exposure to lithium was associated with lack of efficacy or unwanted adverse reactions.
3. Clinical conditions contraindicate the experimental treatment arm (for example thyroid or kidney disease or abnormalities).
4. Pregnant/lactating women.
5. Women of childbearing potential not practicing a reliable method of contraception.

PRIMARY OUTCOME DEFINITION

Suicide completion and acts of deliberate self harm (DSH) will constitute the composite primary outcome. The term "suicide" is defined as an act with a fatal outcome, deliberately initiated and performed by the person with the knowledge or expectation of its fatal outcome.

DSH is defined as intentional self-poisoning or self-injury, irrespective of motivation. Self-poisoning includes the intentional self-ingestion of more than the prescribed amount of any drug, whether or not there is evidence that the act was intended to result in death. This also includes poisoning with non-ingestible substances and gas, overdoses of "recreational drugs" and severe alcohol intoxication where clinical staff consider such cases to be an act of intentional self-harm (rather than recreational binge drinking). Self-injury is defined as any injury that has been intentionally self-inflicted, including self-cutting. The intention to end life may be absent or present to a variable degree. Other terms used to describe this phenomenon are "attempted suicide" and "parasuicide". Some acts of DSH are characterised by high suicidal intent, meticulous planning (including precautions against being found out), and severe lethality of the method used. Other acts of DSH are characterised by no or low intention of suicide, lack of planning and concealing of the act, and low lethality of the method used.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depression (clinical diagnosis, guided by DSM-IV criteria).
* History of attempted suicide or deliberate self-harm in the previous 12 months.
* Inadequate response to at least two antidepressants given sequentially at an adequate dose for an adequate time for the current depressive episode.
* Uncertainty about which treatment arm would be best for participant.
* Age 18 or above.
* Agreement between investigator and patient to enter the study.

Exclusion Criteria:

* In addition to major depression, a primary diagnosis of any concurrent Axis I disorder (according to DSM-IV criteria) will constitute an exclusion criterion; by contrast, any concurrent Axis II disorder (according to DSM-IV criteria) will not constitute an exclusion criterion.
* Previous exposure to lithium was associated with lack of efficacy or unwanted adverse reactions.
* Clinical conditions contraindicate the experimental treatment arm (for example thyroid or kidney disease or abnormalities).
* Pregnant/lactating women.
* Women of childbearing potential not practicing a reliable method of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2009-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Suicide completion and acts of deliberate self harm (DSH) will constitute the composite primary outcome | One year

SECONDARY OUTCOMES:
All-cause mortality | One year
Suicide mortality | One year
Deliberate self-harm or attempted suicide | One year
Change in severity of depressive symptoms from baseline | One year
Adverse reactions during the study | One year

CONTACTS AND LOCATIONS:
Overall Officials: Michele Tansella, MD, Professor of psychiatry, Study Chair — Universita di Verona
Locations (1):
- University of Verona, Verona, Italy

REFERENCES:
- [Derived] Girlanda F, Cipriani A, Agrimi E, Appino MG, Barichello A, Beneduce R, Bighelli I, Bisoffi G, Bisogno A, Bortolaso P, Boso M, Calandra C, Cascone L, Castellazzi M, Corbascio C, Parise VF, Gardellin F, Gennaro D, Hanife B, Lintas C, Lorusso M, Luca A, Luca M, Luchetta C, Lucii C, Maio F, Marsilio A, Mattei C, Moretti D, Nose M, Occhionero G, Papanti D, Pecile D, Percudani M, Prestia D, Purgato M, Restaino F, Romeo S, Sciarma T, Strizzolo S, Tamborini S, Todarello O, Tozzi F, Ziero S, Zotos S, Barbui C. Effectiveness of lithium in subjects with treatment-resistant depression and suicide risk: results and lessons of an underpowered randomised clinical trial. BMC Res Notes. 2014 Oct 17;7:731. doi: 10.1186/1756-0500-7-731. PMID 25326163
- [Derived] Cipriani A, Girlanda F, Agrimi E, Barichello A, Beneduce R, Bighelli I, Bisoffi G, Bisogno A, Bortolaso P, Boso M, Calandra C, Cascone L, Corbascio C, Parise VF, Gardellin F, Gennaro D, Hanife B, Lintas C, Lorusso M, Luchetta C, Lucii C, Cernuto F, Tozzi F, Marsilio A, Maio F, Mattei C, Moretti D, Appino MG, Nose M, Occhionero G, Papanti D, Pecile D, Purgato M, Prestia D, Restaino F, Sciarma T, Ruberto A, Strizzolo S, Tamborini S, Todarello O, Ziero S, Zotos S, Barbui C. Effectiveness of lithium in subjects with treatment-resistant depression and suicide risk: a protocol for a randomised, independent, pragmatic, multicentre, parallel-group, superiority clinical trial. BMC Psychiatry. 2013 Aug 13;13:212. doi: 10.1186/1471-244X-13-212. PMID 23941474